CLINICAL TRIAL: NCT00862433
Title: Vitamin E Pharmacokinetics and Biomarkers in Normal and Obese Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 090097; 09-DK-0097
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12-09

CONDITIONS: Diabetes; Fatty Liver; Obesity; Healthy Volunteers
Keywords: Non-Insulin Dependent Diabetes; Antioxidant; Lipid Peroxidation; Alpha-Tocopherol; Non-Alcoholic Fatty Liver Disease; Health Volunteer; HV; Normal Weight; Overweight; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Fatty Liver; Obesity; Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Overweight | interventions — alpha-Tocopherol; Vitamin E; Ascorbic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): Determine optimal fat content of meal for optimal absorption of vitamin E
  Interventions: Drug: Alpha tocopherol; Other: Vitamin E
- Arm 2 (Experimental): Determine optimal dose of vitamin E.
  Interventions: Drug: Alpha tocopherol; Other: Vitamin E
- Arm 3 (Experimental): Investigate the relationship between vitamin C status and vitamin E turnover
  Interventions: Drug: Alpha tocopherol; Other: Vitamin E; Other: Vitamin C
- NAFLD sub-study (Experimental): Investigate the relationship between fatty liver disease and vitamin E turnover.
  Interventions: Drug: Alpha tocopherol; Other: Vitamin E

INTERVENTIONS:
Drug: Alpha tocopherol — intravenous deuterated vitamin E at doses of 2mg, 5mg, 7.5mg, 10mg and 30mg.
Other: Vitamin E — Deuterated vitamin E, oral and intravenous, at doses of 2mg, 5mg, 7.5mg, 10mg and 30mg.
Other: Vitamin C — Oral vitamin C, one gram daily.
  Arms: Arm 3

SUMMARY:
Background:

* Vitamin E is an antioxidant that reduces the damaging effects of oxygen in the body. Most American men (90%) and women (96%) do not get enough vitamin E from their diets; however, the amount of vitamin E needed by the body has been studied only in men, not women. In addition, it is unknown whether another antioxidant, vitamin C, helps vitamin E in protecting the body. Because vitamin E is a fat-soluble vitamin, how much body fat a person has could affect the amount of vitamin E needed for protection.

Objectives: This study has three arms to examine vitamin E requirements:

* To determine the amount of fat required to get the best vitamin E absorption from a meal.
* To determine the amount (i.e., best dose) of vitamin E that must be consumed before it can be measured in the blood.
* To examine how vitamin E and vitamin C work together in the body, in conjunction with diet and vitamin supplements.

Eligibility:

* Arms 1 and 2: Women between the ages of 18 and 40 years who have a normal weight and body mass index (BMI) of 27 or less.
* Arm 3: Women between the ages of 18 and 40 years who have a normal weight (BMI 27), who are overweight (BMI > 27), or who are overweight (BMI > 27) and have non insulin-dependent diabetes.

Design:

* Arm 1: Five studies, each lasting 1 month with 1 month off between studies (total study = 10 months). Participants will take 500 1,000 mg of vitamin C twice daily for 2 weeks before admission to the clinical center for 1 week.
* Study 1: Participants will eat breakfast containing a known amount of fat, after which they will take a vitamin E pill as well as receive an IV injection of vitamin E. Other foods contain only negligible amounts of vitamin E. Blood and urine samples will measure levels of vitamin E and other substances.
* Studies 2 5: Outpatient visits will consist of the same tests as in Study 1; however, the amount of fat in the breakfast will range from 0% to 40% in random order. During one of the studies, an adipose tissue biopsy will be collected to determine how much vitamin E is in the tissues.
* Arm 2: Five studies, each lasting 1 month with 1 month off between studies (total study = 10 months). Preparation for Arm 2 is the same as in Arm 1. The proportion of fat, muscle, and water in the body will also be measured.
* Study 1: Participants will eat breakfast containing 30% fat, after which they will take a vitamin E pill as well as receive an IV injection of vitamin E. Conditions and procedures are the same as in Arm 1.
* Studies 2 5: Outpatient visits will consist of the same tests as in Study 1; however, the amount of vitamin E in the breakfast will range from 2 to 30 mg in random order.
* Arm 3: Outpatient (2 to 6 weeks) and inpatient studies (4 to 6 weeks).
* Outpatient study: Participants will take 500 1,000 mg of vitamin C daily and provide blood and urine samples, as well as an adipose tissue sample.
* Inpatient studies: Two vitamin E inpatient studies. Before these begin, participants vitamin C blood levels will be reduced by means of a diet low in vitamin C. Blood tests will determine how quickly vitamin C leaves the body. Once the vitamin C level is reduced, the first vitamin E study will begin.

Study A: The procedure for this study is the same as in Arm 2, Study 1.

Study B: The procedure for this study is the same as in Study A, except that the participants blood vitamin C levels will be higher.

DETAILED DESCRIPTION:
Vitamin E (alpha-tocopherol) is essential for humans but determining human dietary requirements has proved difficult. The recommended dietary allowance (RDA) for vitamin E is not met by 96% of American women, without apparent harm. Because vitamin E is an antioxidant, optimum consumption of vitamin E may improve the health of obese women who experience high levels of inflammation and oxidative stress. We hypothesize that vitamin E functions as an antioxidant is related to its tissue stores, and that delivery to tissue stores can be calculated from plasma vitamin E turnover kinetics from slow release pools. We propose turnover kinetics as a new means to estimate vitamin E recommended dietary allowance. We will study vitamin E pharmacokinetics using dual stable-isotope labeled (deuterium) alpha-tocopherols administered orally and intravenously to healthy nonobese, overweight and overweight non-insulin requiring diabetic women. Blood samples will be collected at intervals and vitamin E measured by mass spectrometry. Because ascorbic acid (vitamin C) concentrations may alter alpha-tocopherol pharmacokinetics, subjects will be studied first at low and then high steady state plasma vitamin C concentrations. Before this main study, two preliminary trials will be performed. In preliminary trial 1, fat content for optimal absorption will be assessed because fat-content of a meal may alter vitamin E absorption. The fat content in preliminary trial 1 will be 0 - 40% of calories in the breakfast meal during which vitamin E will be administered. In preliminary trial 2, optimal fat content from preliminary trial 1 will be used, and the vitamin E dose will be varied. Vitamin E dose amount could non-specifically alter vitamin E kinetics. We will therefore determine the largest dose (2-30 mg) that does not non-specifically increase vitamin E turnover, with fat held constant. Additionally, we will measure vitamin E pharmacokinetics as a function of lipid peroxidation biomarkers to provide direct data that can be used to predict vitamin E requirements for women, and to set new recommendations for vitamin E intakes. We will explore new alpha-tocopherol functions, specifically whether gene transcription in human subjects is regulated by vitamin E status in relation to vitamin C status. Because vitamin E turnover may be affected by vitamin C concentrations, we will use a vitamin C depletion-repletion study design to investigate the relationship between vitamin C status and vitamin E turnover.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects to be recruited for the study:

* Healthy women
* Ages 18 to 40 years old
* Able to give informed consent
* Blood pressure <160/90 mm Hg
* Nonobese (BMI less than or equal to 29.9) without diabetes
* Overweight (BMI greater than or equal to 27) without diabetes
* Overweight (BMI greater than or equal to 27) with mild to moderate non-insulin dependent diabetes (Type 2 diabetes)

  * who are treated with diet alone or submaximal doses of oral hypoglycemic agents
  * whose fasting blood sugar is < 200mg/dl or HbA1C < 7.5
  * with no known target organ damage (End organ damage includes the following: proliferative retinopathy, serum creatinine < 1.8 m/dl, ischemic heart disease, congestive heart failure, peripheral vascular disease and peripheral neuropathy)
* No regular medication other than aspirin (other than oral hypoglycemic agents, hormonal contraceptives and medications taken only on an as-needed basis).
* Willingness to use effective contraceptive methods for the duration of the study

EXCLUSION CRITERIA:

Subjects with the following diseases or abnormalities will not be eligible for the study:

* Digestive abnormalities, such as malabsorption or chronic diarrhea
* Organ malfunction, including (but not limited to) liver disease, pulmonary disease, ischemic heart disease, heart failure, stroke, peripheral vascular disease
* Hypertension (blood pressure >160/90)
* Anemia (hematocrit < 30)
* Current or history of serious or chronic illness, including hyperlipidemia or hypercholesterolemia
* Complications from diabetes such as kidney damage (renal insufficiency, serum creatinine >1.8), eye damage (proliferative retinopathy), diabetic neuropathy, coronary artery disease, or peripheral vascular disease
* Tobacco smoking
* Use of medications (other than oral hypoglycemic agents, hormonal contraceptives and medications taken only on an as-needed basis).
* Alcohol or drug abuse
* Insulin treatment
* Pregnancy or lactation (a urine pregnancy test will be performed on all women with reproductive age before each part of the study or monthly as necessary)
* Positive HIV or hepatitis (b or c) screening tests
* Food allergy, to soy or egg, milk protein (casein), or wheat/gluten
* Known coagulopathy
* Unwillingness to use effective contraceptive methods such as barrier methods for the duration of the study.

Patients on antihypertensive medication are excluded even if blood pressure is well controlled because antihypertensive medication may affect vitamin E status, thus introducing a confounding variable. Whether antihypertensive medication interacts with vitamin E is not

known. Patients on insulin treatment are excluded because Insulin treatment indicates a more severe form of diabetes than the mild to moderate type two diabetes that need only dietary treatment or treatment with submaximal doses of oral hypoglycemic agents for adequate blood sugar control. The effect of insulin administration on vitamin E is unknown, and is a confounding factor that will make data interpretation difficult.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10-10 (Actual); Primary Completion 2016-10-21 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Measure Vitamin E Kinetics | q min, hrly, daily
  Fractional vitamin E absorption and rates of plasma vitamin E disappearance after a single dose of oral and intravenous vitamin E

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Levine, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Traber MG, Ramakrishnan R, Kayden HJ. Human plasma vitamin E kinetics demonstrate rapid recycling of plasma RRR-alpha-tocopherol. Proc Natl Acad Sci U S A. 1994 Oct 11;91(21):10005-8. doi: 10.1073/pnas.91.21.10005. PMID 7937827
- [Background] Sowell J, Frei B, Stevens JF. Vitamin C conjugates of genotoxic lipid peroxidation products: structural characterization and detection in human plasma. Proc Natl Acad Sci U S A. 2004 Dec 28;101(52):17964-9. doi: 10.1073/pnas.0408433102. Epub 2004 Dec 17. PMID 15608056 (Retraction: PMID 17724333 Sowell J, Frei B, Stevens JF. Proc Natl Acad Sci U S A. 2007 Sep 4;104(36):14543)
- [Background] Bruno RS, Ramakrishnan R, Montine TJ, Bray TM, Traber MG. alpha-Tocopherol disappearance is faster in cigarette smokers and is inversely related to their ascorbic acid status. Am J Clin Nutr. 2005 Jan;81(1):95-103. doi: 10.1093/ajcn/81.1.95. PMID 15640466
- [Derived] Traber MG, Leonard SW, Ebenuwa I, Violet PC, Niyyati M, Padayatty S, Smith S, Bobe G, Levine M. Vitamin E catabolism in women, as modulated by food and by fat, studied using 2 deuterium-labeled alpha-tocopherols in a 3-phase, nonrandomized crossover study. Am J Clin Nutr. 2021 Jan 4;113(1):92-103. doi: 10.1093/ajcn/nqaa298. PMID 33184629
- [Derived] Violet PC, Ebenuwa IC, Wang Y, Niyyati M, Padayatty SJ, Head B, Wilkins K, Chung S, Thakur V, Ulatowski L, Atkinson J, Ghelfi M, Smith S, Tu H, Bobe G, Liu CY, Herion DW, Shamburek RD, Manor D, Traber MG, Levine M. Vitamin E sequestration by liver fat in humans. JCI Insight. 2020 Jan 16;5(1):e133309. doi: 10.1172/jci.insight.133309. PMID 31821172
- [Derived] Traber MG, Leonard SW, Ebenuwa I, Violet PC, Wang Y, Niyyati M, Padayatty S, Tu H, Courville A, Bernstein S, Choi J, Shamburek R, Smith S, Head B, Bobe G, Ramakrishnan R, Levine M. Vitamin E absorption and kinetics in healthy women, as modulated by food and by fat, studied using 2 deuterium-labeled alpha-tocopherols in a 3-phase crossover design. Am J Clin Nutr. 2019 Nov 1;110(5):1148-1167. doi: 10.1093/ajcn/nqz172. PMID 31495886
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-DK-0097.html